CLINICAL TRIAL: NCT03574649
Title: QUILT-2.024: Phase 2 Neoadjuvant, Consolidation, and Adjuvant Combination NANT Immunotherapy Versus Standard of Care in Subjects With Resectable Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial not initiated
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-2.024
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2018-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Fluorouracil; Cyclophosphamide; DOXO-EMCH; avelumab; ALT-803; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NANT NSCLC Combination Immunotherapy regimen (Experimental)
  Interventions: Drug: Nab-paclitaxel; Drug: Cisplatin; Drug: 5Fluorouracil; Drug: Cyclophosphamide; Biological: ETBX-011; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-4000; Biological: GI-6301; Drug: Aldoxorubicin; Drug: Avelumab; Drug: ALT-803; Biological: haNK
- Standard of Care (Active Comparator)
  Interventions: Drug: Nab-paclitaxel; Drug: Cisplatin; Drug: Docetaxel; Drug: carboplatin

INTERVENTIONS:
Drug: Nab-paclitaxel — 5β,20-Epoxy-1,2α,4,7β,10β,13α-hexahydroxytax-11-en-9-one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)-N-benzoyl-3-phenylisoserine
Drug: Cisplatin — (SP-4-2)-diamminedichloroplatinum(II)
Drug: 5Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
  Arms: NANT NSCLC Combination Immunotherapy regimen
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
  Arms: NANT NSCLC Combination Immunotherapy regimen
Biological: ETBX-011 — adenovirus serotype-5 [Ad5] [E1-, E2b-]-carcinoembryonic antigen [CEA] vaccine
  Arms: NANT NSCLC Combination Immunotherapy regimen
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury vaccine
  Arms: NANT NSCLC Combination Immunotherapy regimen
Biological: ETBX-061 — Ad5 [E1-, E2b-]-mucin 1 [MUC1] vaccine
  Arms: NANT NSCLC Combination Immunotherapy regimen
Biological: GI-4000 — RAS yeast vaccine
  Arms: NANT NSCLC Combination Immunotherapy regimen
Biological: GI-6301 — Brachyury yeast vaccine
  Arms: NANT NSCLC Combination Immunotherapy regimen
Drug: Aldoxorubicin — INNO-206
  Arms: NANT NSCLC Combination Immunotherapy regimen
Drug: Avelumab — Fully human anti-PD-L1 IgG1 lambda monoclonal antibody
  Arms: NANT NSCLC Combination Immunotherapy regimen
Drug: ALT-803 — recombinant human super agonist interleukin-15 (IL-15) complex [also known as IL-15N72D:IL-15RαSu/IgG1 Fc complex]
  Arms: NANT NSCLC Combination Immunotherapy regimen
Biological: haNK — NK-92 [CD16.158V, ER IL-2], Suspension for Intravenous [IV] Infusion (haNK™ for Infusion)
  Arms: NANT NSCLC Combination Immunotherapy regimen
Drug: Docetaxel — Docetaxel
  Arms: Standard of Care
Drug: carboplatin — carboplatin
  Arms: Standard of Care

SUMMARY:
This is a randomized phase 2 study to compare the efficacy of neoadjuvant, consolidation, and adjuvant immunotherapy (NANT NSCLC Combination Immunotherapy; experimental arm) to standard of care (surgery and adjuvant chemotherapy; control arm) in subjects with stage II-IIIa resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically-confirmed stage II-IIIa NSCLC.
4. ECOG performance status of 0 to 2.
5. Have at least 1 measurable lesion of > 1.0 cm.
6. Must have a recent FFPE tumor biopsy specimen following the conclusion of the most recent anticancer treatment and be willing to release the specimen for prospective and exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples prior to the start of treatment on this study for prospective tumor molecular profiling and exploratory analyses.
8. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
9. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, or autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count < 1,000 cells/mm3.
   2. Uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
   3. Platelet count < 75,000 cells/mm3.
   4. Total bilirubin greater than the ULN; unless the subject has documented Gilbert's syndrome).
   5. AST (SGOT) or ALT (SGPT) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. ALP levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   8. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
7. Serious myocardial dysfunction defined by ECHO as absolute LVEF 10% below the institution's lower limit of predicted normal.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for HIV.
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. Participation in an investigational drug study or history of receiving any investigational treatment within 30 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival ( RFS) | 18 months
  time from the date of randomization to the date of first radiographically determined new lesion by RECIST Version 1.1 based on BICR or date of death (by any cause), whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: Undecided